CLINICAL TRIAL: NCT00449618
Title: A Prospective, Randomized, Multi-Center, Double-Blind Crossover Study to Compare Awakening Versus Bedtime Administration of 100 mg Aspirin or Placebo in Subjects With High-Normal Blood Pressure or Mild Essential Hypertension
Brief Title: Comparison of Awakening Versus Bedtime Dosing of Aspirin in Pre-Hypertension or Mild Essential Hypertension
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Not enough recruitment during the proposed period.
Sponsor: University of Vigo (Other)
Collaborators: Hospital Clinico Universitario de Santiago (Other); Bayer (Industry)
Responsible Party: Ramon C. Hermida, University of Vigo
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ASA100-2004/2; 2004-004987-65; 2006-004652-21
Record Dates: First submitted 2007-03-19; First posted 2007-03-20 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2008-12

CONDITIONS: High-Normal Blood Pressure; Mild Essential Hypertension
Keywords: Aspirin; Ambulatory blood pressure monitoring; Chronotherapy; Circadian
MeSH Terms: interventions — Aspirin; Blood Pressure Monitoring, Ambulatory; Chronotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Aspirin 100 mg on awakening
  Interventions: Drug: Aspirin 100 mg; Device: Ambulatory blood pressure monitoring; Procedure: Chronotherapy, timing of medication
- 2 (Active Comparator): Aspirin 100 mg at bedtime
  Interventions: Drug: Aspirin 100 mg; Device: Ambulatory blood pressure monitoring; Procedure: Chronotherapy, timing of medication
- 3 (Placebo Comparator): Placebo on awakening
  Interventions: Device: Ambulatory blood pressure monitoring; Procedure: Chronotherapy, timing of medication; Drug: Placebo
- 4 (Placebo Comparator): Placebo at bedtime
  Interventions: Device: Ambulatory blood pressure monitoring; Procedure: Chronotherapy, timing of medication; Drug: Placebo

INTERVENTIONS:
Drug: Aspirin 100 mg — dose of 100 mg administered on awakening or at bedtime
  Arms: 1; 2
Device: Ambulatory blood pressure monitoring — Blood pressure measured at 20-min intervals from 07:00 to 23:00 hours and at 30-min intervals at night for 48 consecutive hours
Procedure: Chronotherapy, timing of medication — Dosing on awakening versus bedtime
Drug: Placebo — Use of placebo on awakening versus bedtime
  Arms: 3; 4

SUMMARY:
Aspirin (ASA) has been shown to provide marked benefits in the prevention of cardiovascular events, although the potential direct effects of ASA on cardiovascular function remain uncertain. Previous studies have demonstrated that ASA is a potent antioxidative agent that markedly reduces vascular production of superoxide in normotensive and hypertensive rats. In addition, ASA was found to prevent angiotensin II-induced hypertension and cardiovascular hypertrophy, mainly through its antioxidative properties in preventing the generation of superoxide, although ASA apparently did not appear to reduce hypertensive levels of blood pressure (BP). Moreover, recent results have demonstrated that ASA induces nitric oxide (NO) release from vascular endothelium. No attention has been paid, so far, to potential administration time-dependent effects in these studies.

Previous laboratory animal and clinical trial research convincingly demonstrates administration time-dependent (with reference to circadian rhythms) effects of ASA. Thus, the effects of ASA upon lipoperoxides, β-adrenergic receptors, and BP in clinically healthy subjects depend on the circadian timing of ASA administration. Most important, the administration time-dependent influence of ASA on BP was previously demonstrated in a randomized trial on healthy women and in other independent, double-blind, randomized, placebo-controlled clinical trials. The first was conducted on clinically healthy subjects, a second one on normotensive and hypertensive subjects, a third one on pregnant women at high risk for preeclampsia and a fourth one in previously untreated patients with mild hypertension. The findings of these BP studies are consistent; the BP-lowering effect of low-dose ASA is achieved when administered at bedtime but not upon awakening.

In keeping with the chronopharmacological effects of ASA and the previous findings suggesting that ASA at low dose may have a potential beneficial effect on BP, this prospective, randomized, double-blind, crossover study will investigate the potential influence of ASA on BP in subjects with either high-normal BP or diagnosis of mild (grade 1) hypertension. The subjects will receive low-dose ASA or placebo at different times of the day according to their rest-activity cycle, and will be evaluated by 48-hour ambulatory BP monitoring before and after 6 weeks of pharmacologic intervention.

DETAILED DESCRIPTION:
This is a multi-center, prospective, randomized, four-arm, crossover study with double-blind design.

At Visit 1 (week -1) patients will be assessed for eligibility for study participation. Subjects will be advised that study entry cannot be fully determined until the completion of the screening period when all exclusion/inclusion criteria are entirely assessed. Subjects will perform Visit 2 as soon as their laboratory results of Visit 1 are available. At baseline (Visit 2/Day 1), a total of 300 subjects whose eligibility is confirmed will be randomized in a 1:1:1 ratio to one of the treatment groups (aspirin upon awakening, aspirin at bedtime, or placebo--half on awakening, half at bedtime). Subjects will start a first double-blind treatment phase with a total duration of 6 weeks. During this period the subjects will be receiving either aspirin 100 mg or placebo at two different circadian times (either after awakening from nighttime sleep or before bedtime) until the end of this study phase (Visit 3). After this first treatment phase, all subjects will undergo a 2-week wash-out phase with placebo. At Visit 4 (week 8), all subjects will be crossed-over in terms of the circadian time, but keeping their original treatment (either aspirin or placebo), and followed up for a second treatment phase of 6 weeks.

The study duration including all the phases will be 15 weeks.

Safety and efficacy will be assessed at the end of every treatment phase, i.e., at Visits 3 and 5. Safety will also be assessed by phone calls 2 weeks after the initiation of each active treatment phase (weeks 2 and 10). Subjects may be requested to attend the clinic for further evaluation on those weeks if they present any adverse effect.

ELIGIBILITY:
Inclusion Criteria:

* High-normal blood pressure
* Mild essential hypertension

Exclusion Criteria:

* Moderate-severe hypertension.
* Secondary hypertension.
* Grade III/IV hypertensive retinopathy.
* Type 1 diabetes.
* Body mass index ≥ 35 kg/m2
* Cerebrovascular or cardiovascular event during the last 12 months prior to inclusion.
* Pregnant or lactating females.
* History of malignancy within the past five years.
* Shift workers.
* Obstructive sleep apnea.
* Use of disallowed concomitant medication.
* Intolerant to ambulatory BP monitoring (ABPM).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To demonstrate the efficacy of bedtime administration of aspirin by testing the hypothesis of superior 24 hour systolic BP (SBP) lowering compared with either aspirin administered on awakening or with placebo at any circadian time | 14 weeks

SECONDARY OUTCOMES:
To demonstrate that aspirin at bedtime is more effective than aspirin upon awakening and placebo in terms of 24 hour diastolic BP (DBP) lowering | 14 weeks
To demonstrate that aspirin at bedtime is more effective in non-dipper subjects as compared to dippers in terms of nocturnal SBP/DBP lowering, and that this effect is superior to any potential effect on BP of aspirin upon awakening or placebo | 14 weeks
To demonstrate that aspirin at bedtime offers a similar safety profile to aspirin upon awakening and to placebo | 14 weeks
To demonstrate that compliance with aspirin at bedtime is similar to compliance with either aspirin upon awakening or placebo | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ramon C Hermida, Ph.D., Principal Investigator — University of Vigo
Locations (5):
- Spain (5):
  - Centro de Salud de A Guarda, La Guardia, Pontevedra
  - Centro de Salud de Sardoma, Vigo, Pontevedra
  - Centro de Salud de A Doblada, Vigo, Pontevedra
  - C.S. Lérez, Pontevedra
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela